CLINICAL TRIAL: NCT05961020
Title: Effect of Whole-body Vibration on Insulin Resistance in Obese Postmenopausal Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, principle investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p.t.REC\012\004551
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 women was treated by moderate restricted diet for 3 months. (Experimental)
  Interventions: Other: moderate restricted diet
- 20 women treated by whole body vibration. (Experimental)
  Interventions: Device: Total body vibration

INTERVENTIONS:
Device: Total body vibration — Whole-body vibration (WBV) training has been established as a useful method to improve physical fitness in obese individuals. Vibration stimulus during half squatting might suggest a long-term effect of WBV on the endocrine system
  Arms: 20 women treated by whole body vibration.
Other: moderate restricted diet — moderate restricted diet
  Arms: 20 women was treated by moderate restricted diet for 3 months.

SUMMARY:
This study will be conducted to investigate the Effect of whole-body vibration on insulin resistance in obese postmenopausal women

DETAILED DESCRIPTION:
The prevalence of obesity has tripled over the past four decades, imposing an enormous burden on people's health.

Obesity is associated with premature mortality and is a serious public health threat that accounts for a large proportion of the worldwide non-communicable disease burden, including type 2 diabetes, cardiovascular disease, hypertension, and certain cancers.

reported that "Whole-body vibration (WBV) training has been established as a useful method to improve physical fitness in obese individuals. Vibration stimulus during half squatting might suggest a long-term effect of WBV on the endocrine system. Therefore, in this study, The aim to investigate the effect of whole-body vibration on insulin resistance in obese postmenopausal.

ELIGIBILITY:
Inclusion Criteria:

* All women were postmenopausal with no menses at least 1 year.
* Their ages were ranged from 50-60 years old.
* Their body mass index (BMI) > 30 kg/m2.
* They were not engaged in any other treatment program.

Exclusion Criteria:

* Women with body mass index (BMI) < 30 kg/m2.
* Any cardio-respiratory diseases.
* Diabetes mellitus.
* with malignancy.
* with severe hemorrhage, acute viral disease and mental disorders.
* Smokers.
* Women with life threatening disorders as renal failure

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
The Homeostatic model assessment (The HOMA-IR). | up to 3 months
  The Homeostatic model assessment (The HOMA-IR).
  A sample of 5ml of venous blood sample was drawn from all women after 12 hours fasting for measurement of fasting blood glucose, fasting blood insulin and then detection of insulin resistance (by HOMA -IR) through the equation:
  HOMA-IR=(Glucose ×Insulin)/405 glucose in mass unit (mg/dl)
BMI | up to 3 months
  Weight and height were measured to detect the BMI according to the following equation: BMI= weight/height² (Kg/m²)
Waist circumference | up to 3 months
  A non-stretchable tape measurement was used to measure waist circumference for all women in both groups A and B: mid-way between upper border of the lateral iliac crest and the lower border of the lowest rib at the end of gentle expiration with arm relaxed at sides.
Skin fold thickness | up to 3 months
  Skin fold caliper was used to measure skin fold thickness at abdominal region for all women in both groups A and B

CONTACTS AND LOCATIONS:
Locations (1):
- Kerolous Ishak Shehata kelini, Cairo, Egypt